CLINICAL TRIAL: NCT03721211
Title: Imaging With [11C]Martinostat in Breast Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Principal investigator left the study institution.
Sponsor: Christine Elizabeth Edmonds (Other)
Responsible Party: Sponsor-Investigator, Christine Elizabeth Edmonds, Sponsor Investigator, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 17-447
Record Dates: First submitted 2018-10-24; First posted 2018-10-26 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-02

CONDITIONS: Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — martinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [11C]Martinostat (Experimental): * Subjects will be administered [11C]Martinostat, which is synthesized on site at the MGH Martinos Imaging Center
  * All subjects will undergo an MR-PET scan of the thorax, including the breasts, to determine tumor uptake
  * All subjects will be scanned using [11C]Martinostat during an imaging session on a Siemens Biograph mMR integrated MR-PET scanner
  * PET imaging will begin concomitant with radiotracer administration
  Interventions: Drug: [11C]Martinostat; Device: MR-PET scanner

INTERVENTIONS:
Drug: [11C]Martinostat — a type of dye used for radiographic imaging of the HDAC protein
  Other Names: Martinostat
Device: MR-PET scanner — PET, or positron emission tomography, is a type of imaging test that uses a tracer, or dye, to make detailed pictures showing the activities of the cells that make up tissues and organs

SUMMARY:
This research study is studying a PET imaging tracer as a possible means of imaging breast cancer.

The imaging agent involved in this study is:

-[11C]Martinostat (called C-eleven-Martinostat)

DETAILED DESCRIPTION:
This research study is a Pilot Study, which is the first time investigators are examining this study imaging agent in patients who have breast cancer.

The FDA (the U.S. Food and Drug Administration) has approved [11C]Martinostat as an investigational tracer (a type of dye used to for radiographic imaging) in a select few research studies. The FDA has not approved this tracer for any use outside of research.

In this research study, the investigators are investigating the use of a PET tracer called [11C]Martinostat in patients with breast cancer.

The purpose of the study is to take images that can measure the amount of a protein called histone deacetylase, or 'HDAC' in breast tumors. Proteins are molecules made from amino acids that perform activities in the cell for the body to function in a healthy way. Prior research suggests that HDAC levels or amounts can be altered in some breast tumors. The investigators are trying to develop a method of imaging the HDAC protein in breast tumors. This could help them to study protein changes that occur in some breast tumors, and potentially help guide treatment of breast tumors in the future.

In this study, the investigators will take the pictures of the participant's chest, including the breasts, using a PET/MRI scanner. The investigators will the study tracer, or dye, called [11C]Martinostat to make these detailed pictures.

[11C]Martinostat was initially developed to image the HDAC protein within the brain, because amounts or levels of HDAC can be altered in some diseases of the brain. In these previous studies of [11C]Martinostat conducted in humans, there were no adverse events (there have been no problems). While this is not the first time [11C]Martinostat has been used in humans, it is the first study in which the investigators are using this tracer to study breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years or age (required for legal consent)
* Have ECOG performance status ≤2 (Karnofsky ≥60%, see Appendix A)
* Have breast imaging findings from mammogram, ultrasound, or breast MRI that are highly suspicious (i.e. coded as BI RADS 5) for breast cancer.
* Have primary breast tumor that is at least 2 cm in diameter as measured in any dimension on either mammogram, ultrasound, or breast MRI
* Have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

General Exclusion Criteria

* Previously treated breast cancer
* Concurrent malignancy of any type
* Recent breast surgery (within the past 12 months) on the ipsilateral breast as the current breast tumor
* Impaired elimination (as defined as having problems with urination)
* Metallic foreign bodies that would be affected by the MRI magnet, or fear of enclosed spaces likely to make the subject unable to undergo an MRI scan
* Participation in a research study/studies involving radiation exposure within the past 12 months
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, major kidney or liver disease, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnancy
* Currently lactating (either breast feeding or breast pumping)
* Pregnant women are excluded from this study because of the radioactivity of [11C]Martinostat and the resulting risks of teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to administration of [11C]Martinostat, and because lactation may potentially affect the uptake of [11C]Martinostat on PET, breastfeeding women are excluded from the study.

General MR and PET Safety Exclusion Criteria:

* Electrical implants such as cardiac pacemakers or perfusion pumps
* Ferromagnetic implants such as aneurysm clips, surgical clips, prostheses, artificial hearts, valves with steel parts, metal fragments, shrapnel, metallic tattoos anywhere on the body, tattoos near the eye, steel implants, ferromagnetic objects such as jewelry or metal clips in clothing
* Pre-existing medical conditions including a likelihood of developing seizures or claustrophobic reactions, and any greater than normal potential for cardiac arrest
* Inability to lie comfortably on a bed inside a PET camera for 90 minutes as assessed by physical examination and medical history (e.g. back pain, arthritis)
* Pregnancy: A negative serum pregnancy test is required on the day of the PET procedure for female subjects of child-bearing age.
* Body weight of > 250 lbs (weight limit of the MRI table as well as risks to larger patients from MRI elements)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-02-01 (Estimated); Primary Completion 2020-02-28 (Actual); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
PET-MRI Visualization and Quantification of Breast Tumor Uptake of [11C]Martinostat Above Background Uptake, as Assessed by SUV Measurements | up to 2 years
  Evaluate the ability of PET-MRI to visualize and quantify uptake of [11C]Martinostat in breast tumors above background tracer uptake. SUVmax will be collected from the primary breast tumor and the normal background breast tissue. The study is powered to detect a difference in mean background SUVmax of 0.4 in breast parenchyma uninvolved by tumor and breast parenchyma with breast tumor using a two-sample t-test.

SECONDARY OUTCOMES:
Quantitative [11C]Martinostat-PET Uptake in Primary Breast Cancer, and Correlation with Expression of HDAC Isoforms | up to 2 years
  Expression levels of HDAC isoforms will be determined from the baseline breast tumor biopsy specimens via western blot analysis. SUV measurements will be collected from the primary breast tumors on PET-MRI.
Correlation of Total Volume of Distribution of Dynamic [11C]Martinostat Uptake with Expression of HDAC Isoforms | up to 2 years
  Expression levels of HDAC isoforms will be determined from the baseline breast tumor biopsy specimens via western blot analysis. The total volume of [11C]Martinostat distribution will be collected from each PET-MRI.
Comparison of HDAC Isoform Expression by Western Blot Across Breast Tumor Subtypes | up to 2 years
  Expression levels of HDAC isoforms will be determined from the baseline breast tumor biopsy specimens via western blot analysis and will be analyzed for an association with the tumor subtype as determined by expression of the estrogen receptor, progesterone receptor, and HER2 receptor on clinical pathology.
HDAC Expression Levels in Breast Tumors Compared to HDAC Expression in Adjacent Normal Breast Parenchyma | up to 2 years
  Comparison of the expression of HDAC in breast tumors to the expression of HDAC in the adjacent normal breast parenchyma. Expression levels of HDAC isoforms will be determined from the baseline breast tumor biopsy specimens via western blot analysis. Expression of HDAC isoforms in the normal breast parenchyma will be determined from biopsy tissue that is collected from the same breast with the cancer, but in a region of healthy breast parenchyma not involved by tumor.

CONTACTS AND LOCATIONS:
Overall Officials: Christine E Edmond, MD, Study Director — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital Cancer Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No